CLINICAL TRIAL: NCT03204084
Title: Assessment of Low-temperature Plasma Surgery System in Pterygium With Fibrin Glue and Conjunctival Autografts
Status: Completed | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2016011
Record Dates: First submitted 2017-06-19; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Pterygium
Keywords: pterygium,Low temperature plasma
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the LTP group: Patients undergoing pterygium surgery with fibrin glue and conjunctival autografting and receiving Low-temperature Plasma Surgery System(LTP group),
  Interventions: Device: Low-temperature Plasma Surgery System
- the control group: Patients undergoing pterygium surgery with fibrin glue and conjunctival autografting and receiving the conventional method using surgical micro knife and ophthalmic hemostasis(control group)

INTERVENTIONS:
Device: Low-temperature Plasma Surgery System — In pterygium surgery with fibrin glue(FG) and conjunctival autograft we use Low-temperature Plasma Surgery System(LTP)do the ablation of tissue and hemostasis.
  Groups: the LTP group

SUMMARY:
Pterygium is a wing-shaped fibrovascular tissue that has proliferated onto the cornea. Ultraviolet radiation and hot, dusty, windy, dry, smoky environments are regarded as risk factors for pterygium . Surgical removal is the treatment of choice, and surgical wound intraoperative and inflammatory response postoperative have been considered two of the most significant factors that can increase the recurrence rate of pterygium. Low-Temperature Plasma Surgery System(LTP), avoids causing burn injuries to patients, has been introducing into minimally invasive surgery. The mechanism by which this equipment stop bleeding and abolish tissue is to directly occupy the injury with the formed blood clots, plasma flows close the vessel and plasma active particles cause physical and chemical reactions with tissue. The different levels of energy density of plasma can affect the bacteria, cells and cancer cells and even to death, therefore it is widely used in the disinfection of medical devices, dental root canal therapy, skin disease treatment and surgical wound disinfection. Whether it's possible to apply the advantages and benefits of plasma technology in ophthalmic surgery? Like pterygium surgery? However, there is no research to answer until now. In this study, the investigators retrospectively observed the efficacy, postoperative discomfort, inflammation, complications, and recurrence rates in a group of patients for whose LTP was used in pterygium excision and wound hemostasis. The investigators Observe the clinical benefits of LTP in pterygium surgery and find the facilitates and problems it need to be addressed reasonably.

DETAILED DESCRIPTION:
About Plasma It's confirmed that there are 3 physical forms of material existence in human living environment. They are solids, liquids and gass. And any physical form can exist in different states due to the influence of environmental factors. Plasma is the fourth form of material existence. It's composed of ionized conductive gases, including six typical particles, which are electron, positive ion, negative ion, atom or molecule at excited state, atom or molecule at ground state, and photon. Plasma is composed of those positive and negative charged particles and neutral particles, and is a kind of quasi-neutrality gas with collective behavior. It's called plasma when the total negative electric charge equals to the total positive electric charge. 99% visible materials in universe may exist in plasma state, including fixed stars. Plasma can be natural or man-made. For example, the lighting during rainstorms is plasma phenomena, because the high voltage difference between cloud layer and ground makes the air ionized. And neon light and fluorescent lamp are from man-made plasma. The gases in light tube are ionized into plasma state.

About Plasma Low temperature plasma (LTP) Surgery System Low temperature plasma (LTP) Surgery System(made in Chengdu Mechan Electronic Technology Co.,Ltd), which avoids causing burn injuries to patients, has been introducing into minimally invasive surgery. The mechanism by which this equipment stops bleeding is to directly occupy the injury with the formed blood clots, and different from the mechanism of the common electrical hemostatic devices that cauterize the tissues around the bleeding to stem the blood flow. At the same the Plasma Low temperature plasma (LTP) Surgery System has a some biological effects, such as ablation of the organization, this ablation function is generally not penetrating, and only has effect on the contact surface,which can safely handle with the tissue wound and prevent the planting and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* all cases are primary pterygium,a follow-up period of more than 3 months after surgery

Exclusion Criteria:

* no immunorelated disease, ocular surface disease, glaucoma, or eyelid disease. Patients with recurrent pterygium were excluded from the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty-six patients participated in the study. The LTP group consisted of 28 patients (6men) with a mean age±SD of 58.79±1.65 years (range, 42-75 years). The control group consisted of 28 patients (9men) with a mean age±SD of 59.79±1.35 years (range, 41-80years). There were no significant differences in age, gender or eye.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The changes of Best-corrected visual acuity (BCVA), | Before surgery,1-day, 1-week, 1-month, 3-month
  Non-contact ocular pressure measuring instrument

SECONDARY OUTCOMES:
The changes of Patient's subjective discomfort evaluated in terms of the ocular symptom scores(OSS) | Before surgery,1-day, 1-week, 1-month, 3-month
  OSS including five kinds of subjective sensory scale of foreign body sensation, burning sensation, visual fatigue, dryness and eye pain.
conjunctival autograft inflammation | 1-day, 1-week
  Inflammation Grade 0: No dilated corkscrew vessel in the graft Grade 1: 1 bright red, dilated corkscrew vessel crossing the graft-bed margin Grade 2: 2 bright red, dilated corkscrew vessels crossing the graft-bed margin Grade 3: three bright red, dilated corkscrew vessels crossing the graft-bed margin
The changes of the ocular surface inflammation assessed by the Oculus Keratograph○R5M (Oculus Optikgerate GmbH, Wetzlar, Germany), with temporal conjunctival hyperaemia index(TCHI) | Before surgery, 1-week, 1-month, 3-month
  the ocular surface inflammation assessed by the Oculus Keratograph○R5M (Oculus Optikgerate GmbH, Wetzlar, Germany)
The postoperative complications were examined, including dehiscence, dislocation, sclera wound healing defects, granuloma and high intraocular pressure | 1-week, 1-month, 3-month
  Digital slit-lamp photography was performed during each postoperative visit
The recurrence | 3-month
  Digital slit-lamp photography was performed at 3-month
slit-lamp examination | Before surgery,1-week, 1-month
  Corneal epithelium healing
determination of intraocular pressure | Before surgery, 3-month
  Non-contact tonometer
The changes of Patient's subjective discomfort evaluated in terms of the visual analogue scale(VAS) by a questionnaire method | Before surgery,1-day, 1-week, 1-month, 3-month
  Visual Simulation Scoring (VAS): The method is more sensitive and comparable. The specific approach is: on the paper to draw a 10 cm horizontal line, one end of the horizontal line is 0, that painless; the other end is 10, that pain; the middle part of the different degrees of pain. Let the patient according to self-feeling in the horizontal line on a mark, that the degree of pain
The subconjunctival haemorrhage (SCH) | 1-day, 1-week
  Subconjunctival haemorrhage
graft stability according to scoring scale | 1-day, 1-week
  Grade 0: None Grade 1: 25% of the size of the graft Grade 2: 50% of the size of the graft Grade 3: 75% of the size of the graft Grade 4: Haemorrhage involving the entire graft (no subconjunctival vessels visible
  Grade 4: >3 bright red, dilated corkscrew vessels crossing the graft-bed margin Graft stability Grade 0: All four sides of the graft margin are well apposed Grade 1: Gaping/displacement of one side of the graft-bed junction Grade 2: Gaping/displacement of two sides of the graft-bed junction Grade 3: Gaping/displacement of three sides of the graft-bed junction Grade 4: Graft completely displaced from the bed

IPD SHARING:
Plan to Share IPD: Undecided